CLINICAL TRIAL: NCT07174843
Title: An Exploratory Clinical Study to Evaluate the Safety and Efficacy of BZE2204 CD19/CD22/BCMA CAR-T Cells in Subjects With Relapsed or Refractory Active Autoimmune Diseases
Brief Title: An Exploratory Study of CD19/CD22/BCMA CAR-T Cells (BZE2204) in Subjects With Relapsed or Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZE2204-C-01
Record Dates: First submitted 2025-08-19; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Inflammatory Myopathies(IIM); Immune Thrombocytopenia(ITP); Systemic Lupus Erythematosus(SLE)
Keywords: Autoimmune diseases; SLE; IIM; ITP; CAR-T; tri-targets
MeSH Terms: conditions — Myositis; Purpura, Thrombocytopenic, Idiopathic; Lupus Erythematosus, Systemic; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BZE2204 CAR-T cell therapy (Experimental)
  Interventions: Biological: CD19/CD22/BCMA CAR-T cells(BZE2204)

INTERVENTIONS:
Biological: CD19/CD22/BCMA CAR-T cells(BZE2204) — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of BZE2204 CAR T cells.
  On day0 subjects will receive a single dose BZE2204 CAR T cells by intravenous (IV) injection.

SUMMARY:
This is a single arm, open-label, dose escalation and expansion study to evaluate the safety, tolerability and preliminary efficacy of autologous chimeric antigen receptor T (CAR-T) cells targeting CD19/CD22/BCMA(BZE2204) in patients with relapsed or refractory active autoimmune diseases, including idiopathic inflammatory myopathies(IIM), immune thrombocytopenia(ITP), systemic lupus erythematosus(SLE).

DETAILED DESCRIPTION:
This is a single arm, open-label, dose escalation and expansion exploratory study, the primary objective is to evaluate the safety and tolerability of BZE2204 in patients with active relapsed or refractory autoimmune diseases, and determine the maximum tolerated dose (MTD) or recommended dose(RD) for future study. For the secondary objectives, pharmacokinetics(PK), pharmacodynamics (PD) and preliminary will be evaluated.

This study flow comprises of a screening phase( ≤28 days prior to apheresis), apheresis phase (occur upon enrollment, ≤10 days prior to infusion), baseline phase(2-3days before the infusion), BZE2204 CAR-T cells infusion on Day0,safety and efficacy assessments phase (Day1 to Month6), long-term follow-up phase (Month6~Month12).

ELIGIBILITY:
Major Inclusion Criteria:

1. Males or females, aged 18-70 years old
2. Adequate bone marrow, hepatic, renal, coagulation and pulmonary function defined as:

   * Bone marrow reservation: absolute neutrophil count (ANC) ≥1 ×10^9/L; absolute lymphocyte count (ALC)≥ 0.5 ×10^9/L; hemoglobulin ≥80 g/L; platelets ≥50 ×10^9/L(except for ITP);
   * Hepatic function: i: Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 5 upper limit of normal(ULN) (except for elevations are evaluated to be related to autoimmune disease by investigators)and ii: total bilirubin ≤ 2 ULN, (except for Gilbert's syndrome patients, those with total bilirubin ≤ 3 ULN and direct bilirubin ≤ 1.5 ULN can be enrolled).
   * Renal function: serum creatinine ≤ 1.5 ULN , or estimated glomerular filtration rate(eGFR) ≥ 60 mL/min/1.73m2 [eGFR=186×age^-0.203×SCr^-1.154（mg/dl）,female×0.742]
   * Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤1.5 ULN
   * Pulmonary function: Have the minimum level of pulmonary reserve, defined as ≤ CTCAE (Common Terminology Criteria for Adverse Events) grade 1 dyspnea and the SaO2(oxygen saturation)≥ 91% on room air
3. Life expectancy > 6 months
4. Subjects with relapsed or refractory active IIM also need meet following criteria:

   * Subjects with suspected or confirmed dermatomyositis(DM), polymyositis(PM), anti-synthetase syndrome(ASS) and immune-mediated necrotizing myopathy(IMNM, need to be assessed by the investigator that the patient has no safety instability) based on the 2017 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria
   * Positive (+ or above) for at least one myositis-specific antibody (MSA) or myositis-associated antibody (MAA), including anti-TIF-1γ, NXP-2, Mi-2α, Mi-2β, MDA-5, SAE-1/2, SRP, HMGCR, Jo-1, PL-7, PL-12, HA, EJ, OJ, KS, Zo, Tyr, PM-Scl100, PM-Scl75, SSA/Ro-52, SSB/LA, Ku, RNA-PIII, cN1A, etc
   * At screening, the subject must have moderate to severe IIM, defined as manual muscle testing (MMT) ≤ 141 and 2 of the following criteria are met; or CT suggests active interstitial lung disease(ILD)

     1. Physician global activity assessment (PGA) ≥ 2 cm (Visual analogue scale VAS 10 cm);
     2. Patient global activity assessment (PtGA) ≥ 2 cm ( VAS 10 cm scale);
     3. Extramuscular global assessment (Myositis Disease Activity Assessment Tool [MDAAT]) ≥ 2.0 cm (VAS 10 cm scale);
     4. Health assessment questionnaire (HAQ) > 0.25;
     5. Elevation in one or more muscle enzymes (CK, LDH, AST, ALT) is ≥ 1.5 ULN;
   * Lack of efficacy or intolerance to corticosteroids and at least 1 immunosuppressant or biologic agents
5. Subjects with relapsed or refractory active ITP also need meet following criteria

   * Diagnosed with ITP for more than 3 months, including primary ITP and ITP secondary to autoimmune diseases
   * Platelets <50 ×10^9/L with at least twice tests(≥24h interval)
   * At least one platelet glycoprotein specific autoantibody positive
   * Lack of efficacy for first line of therapy, or lack of efficacy/relapse post splenectomy
6. Subjects with relapsed or refractory active SLE also need meet following criteria

   * Diagnosed with SLE according to the 2019 EULAR/ACR classification criteria for at least 6 months
   * Positive autoantibodies: antinuclear antibody (ANA) and/or anti-double strand-DNA(dsDNA) antibody and/or anti-Smith(Sm) antibody
   * SLEDAI-2K scores ≥8 at screening. If the scores for low complement and/or anti-ds-DNA antibody are available, the SLEDAI-2K scores for clinical symptoms (except low complement and/or anti-ds-DNA antibody) should be ≥6
   * Proliferative class III or IV , or class III+V or IV+V lupus nephritis(LN) confirmed by biopsies within 12 months; urine protein > 1.0g/24h or urine protein creatinine ratio (UPCR) >1000mg/g and PGA>1
   * Lack of efficacy or intolerance to at least one immunosuppressant and/or one biologic in medical history; for LN patients, relapse during maintenance post induction therapy is also eligible.

Major Exclusion Criteria:

1. A history of severe hypersensitivity or allergic reactions, or contraindications or hypersensitivity to any component of the investigational drug
2. Presence of any serious heart diseases defined in the protocol
3. A medical history of severe central nervous system or symptoms within 6 months
4. Any concurrent malignancy or a history of malignancy with exceptions indicated in the protocol
5. Clinically significant hemorrhage symptoms or definite bleeding tendencies (except for events caused by ITP) within 6 months prior to screening; arteriovenous thrombosis events within 6 months prior to screening
6. Any positive results of contagious diseases as following:

   * Human immunodeficiency virus (HIV) antibody positive;
   * HBsAg positive; or HBcAb/HBeAb positive (subjects with HBV DNA copy numbers below the lower limit of detection can be enrolled);
   * hepatitis C antibody (HCV-Ab) positive (the subjects with HCV RNA below the lower limit of detection can be enrolled) or a known medical history of hepatitis C;
   * Treponema pallidum antibody (TP-Ab) positive
   * Epstein-Barr virus(EBV), cytomegalovirus(CMV) antibody positive and copy number is above the limit
7. Active tuberculosis or latent tuberculosis that has not been adequately treated
8. Evidenced viral, bacterial or fungal infection that is uncontrolled or requires systemic antimicrobial therapy
9. Requirements of wash-out period for specific treatment are not met(detailed in protocol)
10. Subjects with relapsed or refractory active IIM will be excluded in the following situations:

    * Inclusion body myositis, amyopathic dermatomyositis or secondary myositis with documented medical history
    * Severe muscle damage
    * Uncontrolled extra muscle damage relating to PM or DM
11. Subjects with relapsed or refractory active ITP will be excluded if platelet < 10x10^9/L with active bleeding or bleeding score ≥5
12. Subjects with relapsed or refractory active SLE will be excluded if the subject has lupus crisis within 3 month, active CNS lupus, severe hemolytic anemia, severe thrombocytopenic purpura etc
13. Any situations evaluated by investigators that may prevent the subjects from participating in the study, or may confound the study results, or participation in this study is not in the best interests of the subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The frequency and severity of adverse events(AE) and serious adverse events(SAE) | From leukapheresis to 6 months post CAR-T infusion
The frequency of dose-limiting toxicity(DLT) | Day0 to Day28

SECONDARY OUTCOMES:
Chimeric antigen receptor T cell (CAR-T) levels in peripheral blood at each time point. | Day0-Month6 post infusion
Chimeric antigen receptor transgene levels in peripheral blood at each time point | Day0-Month6 post infusion
Cytokines levels of IL-2(interleukin), IL-4, IL-6,IL-8, IL-10, IL-12p70, IL-13, IL-1β, TNF-a, IFN-r in peripheral blood at each time point. | Day-3 to Month6 post infusion
B cell levels in peripheral blood at each time point | Day-3 to Month6 post infusion
Immunoglobulins in peripheral blood at each time point | Day-3 to Month6 post infusion
The level of muscle enzymes AST(aspartate transaminase), ALT(alanine transaminase), LDH(lactate dehydrogenase), CK(creatine kinase) in peripheral blood at each time point in idiopathic inflammatory myopathies (IIM) | Day-3 to Month6 post infusion
The time of stopping steroids, immunosuppressants for autoimmune disease post infusion | Day0-Month6 post infusion
The proportion of subjects with idiopathic inflammatory myopathies(IIM) achieving 2016 total improvement score(TIS) mild, moderate, major improvement; the time to the improvement and the duration of improvement. | Month3, Month6
The proportion of subjects with immune thrombocytopenia(ITP) achieving complete remission | Month3, Month6
The proportion of subjects with immune thrombocytopenia(ITP) achieving partial remission | Month3, Month6
The proportion of subjects with systemic lupus erythematosus(SLE) achieving SLE Responder Index-4(SRI-4); the time to response and the duration of the response | Month3, Month6
The change of SLE Disease Activity Index 2000(SLEDAI-2K) post infusion | Month3, Month6

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mengchao Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No